CLINICAL TRIAL: NCT03175627
Title: Clinical Investigation Of A Bulk Fill Composite In Class II Restorations In Adult Subjects
Brief Title: Clinical Performance of Posterior Composite Tooth Fillings in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Adriana Cordero Wilson, Clinical Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-050008
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Dental Caries; Dental Restoration Failure
Keywords: Dental caries; Proximal surfaces; Posterior teeth; Carious lesions; Tooth diseases; Dental restorations; Composite resin
MeSH Terms: conditions — Dental Caries; Tooth Diseases

STUDY DESIGN:
Intervention Model Description: In a split-mouth design, each participant will receive 2 matched restorations, one of each material.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind (Subject, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Filtek One (Active Comparator): Bulk fill composite material used for posterior tooth fillings.
  Interventions: Device: Filtek One
- Filtek Z250 (Active Comparator): Composite material used for incremental filling of posterior teeth.
  Interventions: Device: Filtek Z250

INTERVENTIONS:
Device: Filtek One — Restoring a posterior permanent tooth in need of a filling applying Filtek One using bulk fill technique.
  Other Names: 3M™ Filtek™ One Bulk Fill Restorative
  Arms: Filtek One
Device: Filtek Z250 — Restoring a posterior permanent tooth in need of a filling applying Filtek Z250 using incremental filling technique.
  Other Names: 3M™ Filtek™ Z250 Universal Restorative
  Arms: Filtek Z250

SUMMARY:
The purpose of this study is to determine whether a new tooth-colored composite material is effective for load-bearing dental fillings.

DETAILED DESCRIPTION:
In this post-market prospective randomized controlled clinical trial, posterior class II restorations will be evaluated for their clinical performance. The study will investigate the survival and efficacy of a bulk-filled composite resin restorative material for a period of 2 years. The bulk fill composite will be used according to indication and applied in approximal two- or three-surface restorations in permanent teeth.

ELIGIBILITY:
Inclusion Criteria:

* be older than 18 years of age
* have 2 back teeth with similar size tooth decay or failed fillings, that are in need of new moderate-size fillings
* both study teeth must be vital (tested with cold)
* both study fillings must be visible on the cheek-side of the tooth.

Exclusion Criteria:

* do not meet all inclusion criteria
* are under active orthodontic treatment
* have severe medical complications
* have dry mouth
* have chronic gum disease or poor oral hygiene
* are unavailable for long term recall (minimum of 2 years required)
* cannot tolerate the rubber dam
* have an unstable tooth contacts
* have severe bruxing or clenching, or are in need of jaw joint therapy
* are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with restoration failure of either material | 2 years
  Restoration failure is based on clinical performance criteria according to the Fédération Dentaire Internationale (FDI) rating system. An assessment of score 5, indicating poor performance, in any of the three categories esthetic, functional or biological performance will be considered a failure.

SECONDARY OUTCOMES:
Clinical performance score for each restoration | 2 years
  Quality rating for each restoration/material based on the FDI clinical performance scores (1-5) for the three categories esthetic, functional and biological performance.
Confirmation of material safety | 2 years
  Number of participants with unanticipated treatment-related Adverse Events as assessed by • Fatal, • Persistent disability or significant incapacity, • Congenital anomaly/birth defect or cancer, • Life-Threatening, • Associated with overdose, • Required hospital admission or prolongation of hospitalization (Adverse Events Reporting Requirements LSUHSC-NO IRB).

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde C Peters, DMD, PhD, Study Director — LSUHSC School of Dentistry
Locations (1):
- Lousiana State University Health Science Center, School of DentistrySchool of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No